CLINICAL TRIAL: NCT00544284
Title: A Phase I Study of Bortezomib and Temozolomide in Patients With Refractory Solid Tumors
Brief Title: Bortezomib and Temozolomide in Treating Patients With Brain Tumors or Other Solid Tumors That Have Not Responded to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04032; P30CA033572 (NIH); CHNMC-04032; CDR0000570245 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; recurrent adult brain tumor; adult gliosarcoma; adult mixed glioma; adult anaplastic oligodendroglioma; primary central nervous system lymphoma; adult diffuse astrocytoma; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic meningioma; adult melanocytic lesion; adult meningeal hemangiopericytoma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult papillary meningioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma; tumors metastatic to brain; unspecified adult solid tumor, protocol specific; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neoplasm Metastasis; Glioblastoma; Astrocytoma; Brain Neoplasms; Gliosarcoma; Glioma; Oligodendroglioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Glioma, Subependymal; Meningioma; Pinealoma | interventions — Bortezomib; Temozolomide

ARMS (1):
- Treatment (temozolomide, bortezomib) (Experimental): GROUP A: Patients receive oral temozolomide once a day on days 1-5 and bortezomib IV on days 2, 5, 9, and 12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. GROUP B: Patients receive temozolomide and bortezomib as in group A. Cohorts of patients in both groups receive escalating doses of both study drugs until the maximum tolerated doses are determined. All patients undergo blood sample collection periodically for pharmacokinetic studies. Samples are analyzed for bortezomib concentration (groups A and B) and trough levels of anticonvulsants (group A only).
  Interventions: Drug: bortezomib; Drug: temozolomide; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib
Drug: temozolomide
Other: pharmacological study

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with temozolomide in treating patients with brain tumors or other solid tumors that have not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose-limiting toxicities and maximum tolerated doses of bortezomib and temozolomide in patients with recurrent high-grade gliomas, recurrent metastatic brain tumors, or other refractory solid tumors.

Secondary

* To evaluate the pharmacokinetics of bortezomib in patients taking hepatic enzyme-inducing anticonvulsants (Group A) and in those who are not (Group B).
* To describe the proportion of study patients treated with bortezomib and temozolomide who obtain a confirmed complete response or partial response.
* To report the percentage of patients with 6-month progression-free survival.

OUTLINE: Patients are stratified according to concurrent hepatic enzyme-inducing anticonvulsants (HEIAs) (Group A) versus concurrent anticonvulsant drugs that cause modest or no induction of hepatic metabolic enzymes OR no anticonvulsant drugs (Group B).

* Group A: Patients receive oral temozolomide once a day on days 1-5 and bortezomib IV on days 2, 5, 9, and 12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Group B: Patients receive temozolomide and bortezomib as in group A. Cohorts of patients in both groups receive escalating doses of both study drugs until the maximum tolerated doses are determined.

All patients undergo blood sample collection periodically for pharmacokinetic studies. Samples are analyzed for bortezomib concentration (groups A and B) and trough levels of anticonvulsants (group A only).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumors including the following

  * Recurrent high-grade glioma
  * Recurrent metastatic brain tumors
  * Recurrent primary brain tumor including primary CNS lymphoma
  * Other refractory solid tumors
* Unresectable disease for which standard curative or palliative measures do not exist or are no longer effective
* Measurable or nonmeasurable disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 mg/dL
* AST ≤ 4.0 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patient must be able to understand and is willing to sign a written informed consent document

Exclusion criteria:

* Any of the following conditions:

  * Myocardial infarction within the past 6 months or New York Heart Association class III or IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * ECG evidence of acute ischemia or active conduction system abnormalities

    * Any ECG abnormalities prior to study entry must be documented by the investigator as not medically relevant
* Serious medical or psychiatric illness that would, in the opinion of the investigator, potentially interfere with the completion of treatment
* History of sensitivity to boron or mannitol

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea-containing chemotherapy), immunotherapy, or radiotherapy and recovered
* More than 10 days since prior anticonvulsant drugs that induce hepatic metabolic enzymes for patients in group A
* Recovered from major surgery

  * Corticosteroids for cerebral edema allowed provided the patient is on a stable dose for at least 1 week

Exclusion criteria:

* Patients enrolled on another clinical trial
* HIV-positive patients on antiretroviral therapy
* Concurrent chemotherapy or radiotherapy
* Patient requires anti-seizure medication but is not on a stable dose and agent of anti-seizure medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics | Day 9
Confirmed complete or partial response | 6 months
Percentage of patients with 6-month progression-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

REFERENCES:
- [Derived] Portnow J, Frankel P, Koehler S, Twardowski P, Shibata S, Martel C, Morgan R, Cristea M, Chow W, Lim D, Chung V, Reckamp K, Leong L, Synold TW. A phase I study of bortezomib and temozolomide in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2012 Feb;69(2):505-14. doi: 10.1007/s00280-011-1721-x. Epub 2011 Aug 18. PMID 21850464